CLINICAL TRIAL: NCT00930072
Title: Safety and Efficacy of Cervical Sympathetic Block in Patients With Cerebral Vasospasm Following Aneurysmal Subarachnoid Hemorrhage - Pilot Study
Brief Title: Safety Study of Cervical Sympathetic Block for Cerebral Vasospasm Following Aneurysmal Subarachnoid Hemorrhage
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor Enrollment
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Miriam Treggiari, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34225
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Vasospasm
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Block (Experimental)
  Interventions: Drug: Cervical Sympathetic Block (bupivicaine, clonidine)
- Standard Care (No Intervention)

INTERVENTIONS:
Drug: Cervical Sympathetic Block (bupivicaine, clonidine) — 12-15ml solution of bupivicaine .5% containing 50 mcg of clonidine for cervical sympathetic block administered in a single injection.
  Other Names: Bupivicaine; Clonidine
  Arms: Block

SUMMARY:
To evaluate the feasibility of performing a cervical sympathetic block in patients with severe cerebral vasospasm involving the anterior cerebral circulation following aneurysmal SAH.

ELIGIBILITY:
Inclusion Criteria:

1. High grade spontaneous SAH (Fisher Grade III and IV)
2. Secured aneurysm (clipped/coiled)
3. Evidence of severe vasospasm - MCA mean flow velocity >200 cm/sec and Lindegaard ratio >6 OR Symptomatic vasospasm with either angiographic evidence (no angioplasty), or at least moderate severity according to TCD criteria (MCA mean flow velocity >150 cm/sec and Lindegaard ratio >3, or ACA vasospasm)
4. Age ≥18

Exclusion Criteria:

1. Allergy to local anesthetic or contrast
2. Coagulation disorders with PT <70%, or INR >1.4, or PTT >1.5 times control and/or platelets <70,000x106/L
3. Use of enoxaparin within 12 hours
4. Use of clopidogrel within 7 days
5. Use of coumadin within 5 days
6. Use of ticlopidine within 14 days
7. Use of intravenous thrombolytics within 10 days
8. Any use of hirudin derivatives during ICU stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of performing a cervical sympathetic block in patients with severe cerebral vasospasm involving the anterior cerebral circulation following aneurysmal SAH. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Treggiari, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No